CLINICAL TRIAL: NCT02042885
Title: A Two-part Phase 1/2a, Open-label, Dose Escalation Study to Evaluate the Tolerability and Preliminary Antitumour Activity of OPB-111001 in Patients With Advanced Cancers That Are Poorly Responsive to Standard Anticancer Treatment
Brief Title: A Clinical Trial to Determine the Most Suitable Dose of OPB-111001 in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Novel Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 314-12-401; 2013-001249-15 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer; Salivary Gland Cancer; Endometrial Cancer; Squamous Cell Carcinoma of the Cervix; Breast Cancer; Ovarian Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Neoplasms; Endometrial Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Regimen A Escalation (Experimental): 1: OPB-111001, orally, once weekly
  Interventions: Drug: OPB-111001
- 2: Regimen A Extension (Experimental): 2: OPB-111001, orally, once weekly
  Interventions: Drug: OPB-111001
- 3: Regimen B Escalation (Experimental): 3: OPB-111001, orally, 2 - 3 times per week
  Interventions: Drug: OPB-111001
- 4: Regimen B Extension (Experimental): 4: OPB-111001, orally, 2 - 3 times per week
  Interventions: Drug: OPB-111001

INTERVENTIONS:
Drug: OPB-111001

SUMMARY:
The purpose of this study is to determine the tolerability profile of OPB-111001 and to determine the most suitable dose of OPB-111001 in patients with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patients with prostate cancer that is recurrent or did not respond to previous hormone therapy and/or who have exhausted standard treatment options.

For the dose escalation parts only:

Patients who have exhausted standard treatment options with recurrent or refractory cancer (ovarian cancer, cervical squamous cell carcinoma, breast cancer, salivary gland cancer, endometrial cancer)

* Histologically or cytologically documented diagnosis of cancer
* Measurable disease according to RECIST Version 1.1 or for prostate cancer also evaluable disease according to Prostate Cancer Working Group 2 (PCWG2) eligibility criteria or for ovarian cancer also evaluable disease (non-measurable) according to Gynaecologic Cancer Intergroup (GCIG) criteria
* Absolute neutrophil count ≥1.5 (1500/mm3) and platelets ≥100 × 109/L (without platelet transfusion within the last 4 weeks before first study drug administration), and haemoglobin ≥9 g/dL at Screening
* Alanine aminotransferase and aspartate aminotransferase ≤2.5 × the upper limit of normal (ULN), Total bilirubin ≤1.5 × ULN (exception: patients with liver metastasis are allowed to have aspartate aminotransferase ≤5 × ULN and alanine aminotransferase ≤5 × ULN) at screening
* Albumin ≥26 g/L at Screening

Exclusion Criteria:

* Concurrent prior treatment-related toxicity of Grade 2 or higher. Exception: any toxicity that is in the view of the investigator not a clinically significant safety risk for Investigational medicinal product (IMP) administration.
* Previous treatment with cytotoxic chemotherapy or other anticancer therapy within 4 weeks before the first dosing with study drug (at least 6 weeks for mitoxantrone, nitrosurea, and bicalutamide).
* Treatment with systemic glucocorticosteroids of more than a 2 mg dexamethasone equivalent per day or in cases of treatment with ≤2 mg dexamethasone equivalent per day:

  1. Dosing was changed within 6 weeks before Screening or
  2. The patient's cancer is responding to glucocorticosteroid intake
* Radiation therapy within 4 weeks prior to the first dosing with IMP.
* Treatment with a systemic IMP in a clinical trial within 28 days before the Screening Visit.
* Current or past history of clinically significant gastrointestinal disease or major gastrointestinal surgery, malabsorption syndrome, or other conditions that could interfere with enteral absorption.
* Concurrent clinically significant unrelated systemic illness (e.g., serious infection) or significant pulmonary, hepatic, or other organ dysfunction that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose / Recommended Phase 2 dose; Tolerability | after 2 or 6 weeks depending on study part; continously

SECONDARY OUTCOMES:
Pharmacokinetic parameters for OPB-111001 and its metabolites | repeatedly until end of study (average of 3 months assumed)
  Frequent sampling during Cycle 1 to 3, D1 only from Cycle 4 onwards
Assessment of antitumor activity as defined by Response Evaluation Criteria in Solid Tumours (RECIST) | repeatedly every 8th week until end of study (average of 3 months assumed)
Prostate-specific antigen (PSA) response in patients with prostate cancer | repeatedly (Cycle 1 to 3 on Day 1, then every 4th week) until end of study (average of 3 months assumed)
Cancer antigen 125 (CA 125) response in patients with ovarian cancer | repeatedly (Cycle 1 to 3 on Day 1, then every 4th week) until end of study (average of 3 months assumed)
Time to treatment failure | At end of study (after average of 3 months assumed)

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, Prof. Dr., Principal Investigator — The Institute of Cancer Research, Royal Marsden NHS Foundation Trust London United Kingdom; Sarah Blagden, Dr., Principal Investigator — NIHR/Wellcome Trust Imperial CRF, Imperial College Healthcare NHS Trust, Imperial Center for Translational and Experimental Medicine (L-Block), Hammersmith Hospital London, United Kingdom
Locations (2):
- United Kingdom (2):
  - The Institute of Cancer Research, Royal Marsden NHS Foundation Trust, London, Sutton, Surrey
  - NIHR/Wellcome Trust Imperial CRF/Imperial College Healthcare NHS Trust, Imperial Centre for Translational and Experimental Medicine (L-Block), Hammersmith Hospital, London